CLINICAL TRIAL: NCT01900015
Title: Changes in Liver Steatosis After Switching From Efavirenz to Raltegravir Among HIV/HCV-Coinfected Patients Receiving Two Nucleoside Analogs Plus Efavirenz: The Steral Study
Brief Title: Changes in Liver Steatosis After Switching to Raltegravir in HIV/HCV Coinfection
Acronym: STERAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan Macías (Other Government)
Responsible Party: Sponsor-Investigator, Juan Macías, PhD, Andaluz Health Service
Organization: Andaluz Health Service (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STERAL/50410
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: HCV Coinfection; HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Active Comparator): Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.
  Interventions: Drug: Raltegravir
- Efavirenz (Active Comparator): Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Raltegravir — Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.
  Other Names: Issentres
  Arms: Raltegravir
Drug: Efavirenz — Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.
  Other Names: Sustiva
  Arms: Efavirenz

SUMMARY:
Primary Objective:

To compare the impact of switching from efavirenz (EFV) plus two nucleoside analogs to rategravir (RAL) plus two nucleoside analogs versus keeping the same antiretroviral regimen on hepatic steatosis (HS) as measured by the controlled attenuation parameter (CAP) among HIV/HCV-coinfected patient.

Secondary Trial Objective:

1. To compare the proportion of HIV/HCV-coinfected patients with one category decrease in the grade of HS between patients continuing with EFV plus two nucleoside analogs and those switching from EFV plus two nucleoside analogs to RAL plus two nucleoside analogs.
2. To evaluate the proportion of patients who maintain viral control (HIV RNA < 50 copies/mL) after switching.

Design:

Open-label, randomized clinical trial to evaluate safety (phase IV)

Condition:

HIV and HCV coinfection.

Intervention:

Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.

DETAILED DESCRIPTION:
Primary Objective:

To compare the impact of switching from efavirenz (EFV) plus two nucleoside analogs to rategravir (RAL) plus two nucleoside analogs versus keeping the same antiretroviral regimen on hepatic steatosis (HS) as measured by the controlled attenuation parameter (CAP) among HIV/HCV-coinfected patient.

Secondary Trial Objective:

1. To compare the proportion of HIV/HCV-coinfected patients with one category decrease in the grade of HS between patients continuing with EFV plus two nucleoside analogs and those switching from EFV plus two nucleoside analogs to RAL plus two nucleoside analogs.
2. To evaluate the proportion of patients who maintain viral control (HIV RNA < 50 copies/mL) after switching.

Design:

Open-label, randomized clinical trial to evaluate safety (phase IV)

Condition:

HIV and HCV coinfection.

Intervention:

Patients on current EFV plus two nucleoside analogs will be randomly assigned to switch EFV to RAL (400mg BID), maintaining nucleoside analogs unchanged, or to continue the current regimen.

Study population and sample size HIV-infected patients with concomitant coinfection by HCV, as shown by detectable plasma HCV RNA, not candidates for therapy against HCV infection during the 48 week period of the Number of patients to recruit: 96, 48 patients per treatment group should be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must be willing and able to provide written informed consent for the trial.
2. Each subject must be ≥ 18 years of age.
3. Each subject must be male or non-pregnant, non-breastfeeding female
4. Each subject must have diagnosis of HIV infection.
5. Each subject must have concomitant coinfection by HCV as shown by detectable plasma HCV RNA.
6. Each subject must have stable treatment with EFV plus two nucleoside analogs for ≥24 weeks.
7. Each subject must have at least 2 documented plasma HIV RNA <50 copies/ml during the last 24 weeks, as observed in, at least, two clinical visits.
8. Each subject must have HS involving more than 10% of hepatocytes, as determined by a CAP measurement ≥238 dB/m.
9. Each sexually active female subject of child-bearing potential must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 3 months after stopping the medication.Medically accepted methods of contraception include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed IUD, inert or copper-containing IUD, hormone releasing IUD, systemic hormonal contraceptive, and surgical sterilization (eg,hysterectomy or tubal ligation).Postmenopausal women are not required to use contraception.Postmenopausal is defined as at least 12 consecutive months without a spontaneous menstrual period.
10. Each sexually active male subject with a female partner(s) of child-bearing potential must also provide written informed consent to provide information regarding any pregnancy.
11. Average daily alcohol intake lower than 50 g for men and 40 g for women.

Exclusion Criteria:

1. The subject has an allergy/sensitivity to investigational product or its/their excipients.
2. The female subject is nursing.
3. The female subject is pregnant or intending to become pregnant.
4. History of ARV failure or documented resistance.
5. Baseline resistance to EFV or to any of the nucleoside analogues inhibitors in the regimen.
6. The subject has any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the trial evaluations or optimal participation in the trial.
7. The subject has active AIDS-defining event (CDC-C) within 24 weeks before screening.
8. The subject is candidate for therapy against HCV infection during the 48 week trial period in the opinion of the investigator.
9. The subject has a history of malignant neoplasia.
10. Active illicit drug use or any other condition that may compromise the study drug adherence in the opinion of the investigators.
11. The subject has used any investigational drugs within 30 days of Baseline.
12. A subject who has participated in any other clinical trial within 30 days,inclusive, of signing the informed consent form of the current trial.
13. The subject or a family member is among the personnel of the investigational or SPONSOR staff directly involved with this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
To compare the impact of switching from EFV plus two nucleoside analogs to RAL plus two nucleoside analogs versus keeping the same antiretroviral regimen on HS as measured by CAP among HIV/HCV-coinfected patients. | 48 weeks

SECONDARY OUTCOMES:
To evaluate the proportion of patients who maintain viral control (HIV RNA < 50 copies/mL) after switching. | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Macías, MD, PhD, Principal Investigator — Infectious Diseases and Microbiology Unit. Hospital Universitario de Valme. Servicio Andaluz de Salud
Locations (10):
- Spain (10):
  - Hospital La Línea, La Línea de la Concepción, Cádiz
  - H.U. Valme, Seville, Seville
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Infanta Elena, Huelva
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macias J, Mancebo M, Merino D, Tellez F, Montes-Ramirez ML, Pulido F, Rivero-Juarez A, Raffo M, Perez-Perez M, Merchante N, Cotarelo M, Pineda JA; Spanish AIDS Research Network-HEP09 Study Group. Changes in Liver Steatosis After Switching From Efavirenz to Raltegravir Among Human Immunodeficiency Virus-Infected Patients With Nonalcoholic Fatty Liver Disease. Clin Infect Dis. 2017 Sep 15;65(6):1012-1019. doi: 10.1093/cid/cix467. PMID 28903510
- See also: Abstract presented at CROI 2017. Poster available to download — http://www.croiconference.org/sessions/changes-liver-steatosis-after-switching-efavirenz-raltegravir-steral-study-0
- See also: CROI webcast. THEMED DISCUSSION: OBESITY AND FATTY LIVER DISEASE — http://www.croiwebcasts.org/p/2017croi/croi33405